CLINICAL TRIAL: NCT06487286
Title: Levels of Visfatin/NAMPT in Human Milk.VISFAMILK
Brief Title: Levels of Visfatin/NAMPT in Human Milk
Acronym: VISFAMILK
Status: Recruiting | Type: Observational
Sponsor: Paolo Manzoni Study Group (Other)
Collaborators: Università degli Studi del Piemonte Orientale Amedeo Avogadro (Other)
Responsible Party: Sponsor-Investigator, Paolo Manzoni Study Group, Principal Investigator, Head of Department of Maternal, Neonatal and Infant Medicine, Associate Professor, Paolo Manzoni
Organization: Paolo Manzoni (Other)
Other Study IDs: 4
Record Dates: First submitted 2024-06-27; First posted 2024-07-05 (Actual); Last update posted 2024-11-14 (Actual); Status verified 2024-11

CONDITIONS: Visfatin Levels in Maternal Milk Samples; Birth Weight
Keywords: Newborns; Visfatin; Breastfeeding
MeSH Terms: conditions — Birth Weight; Breast Feeding | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: observational study — observational study

SUMMARY:
Visfatin, released in maternal milk at different concentrations related to the maternal conditions, could act as a biomarker with a prognostic/predictive value to determine different newborn clinical conditions, particularly the weight loss of the neonate.

DETAILED DESCRIPTION:
The aim of the study is to analyse a retrospective cohort of well characterized mothers in their post-partum period, and to measure Visfatin levels through collection of maternal milk samples. They will be collected in three different moments after the birth (48 hours, 7 days and 30 days) and Visfatin levels will be analysed through an ELISA kit Adipogen. In parallel, the levels of Visfatin will be evaluated in the maternal plasma/serum collected after 1-2 days postpartum.

Lastly, correlations between Visfatin levels and biological/clinical features of mothers and newborns will be explored.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female infants born after 37 weeks' gestation who do not have conditions related to congenital abnormalities
* Maternal hospitalization
* Acquisition of the informed consent form signed by the patient

Exclusion Criteria:

* Refusal of the patient to participate in the study
* Presence of hypogalactia or agalactia in the patient

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: 30 women, hospitalized after childbirth, with respective healthy, breastfed infants
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2024-10-24 (Actual); Primary Completion 2025-04-23 (Estimated); Study Completion 2025-04-23 (Estimated)

PRIMARY OUTCOMES:
Visfatin levels | 48 hours, 7 days and 30 days
  Visfatin levels in maternal milk samples
Visfatin levels | 1-2 days post-partum
  Visfatin levels in maternal plasma/serum

SECONDARY OUTCOMES:
values of Visfatin | 6 months
  correlate the values of Visfatin to different demographic and clinical characteristics of the lactating mothers
values of Visfatin | 6 months
  correlate the values of Visfatin to different biological/clinical features of the newborns; in particular, we will focus attention on the weight loss of the neonate

CONTACTS AND LOCATIONS:
Locations (1):
- Ospedale degli Infermi - ASL BI, Ponderano, BI, Italy